CLINICAL TRIAL: NCT01564979
Title: Effect on Tear Functions of Pretarsal and Preseptal Techniques of Botulinum Toxin Type A Injection in Hemifacial Spasm
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, kitthisak kitthaweesin, Assoc Prof, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KTS-001-BTX
Record Dates: First submitted 2012-03-18; First posted 2012-03-28 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Hemifacial Spasm
Keywords: botulinum toxin; facial nerve; hemifacial spasm; tears
MeSH Terms: conditions — Hemifacial Spasm; Lacerations | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- preseptal (Experimental)
  Interventions: Drug: preseptal injection of botulinum toxin type A
- pretarsal (Experimental)
  Interventions: Drug: pretarsal injection of Botulinum toxin type A

INTERVENTIONS:
Drug: preseptal injection of botulinum toxin type A — botulinum toxin type A (Botox)2.5 units, 5 points
  Other Names: Botox
  Arms: preseptal
Drug: pretarsal injection of Botulinum toxin type A — Botulinum toxin type A 2,5 units, 5 points
  Other Names: Botox
  Arms: pretarsal

SUMMARY:
The purpose of this study is to determine whether pretarsal and preseptal techniques of Botulinum toxin type A injection have any effect on tear functions.

DETAILED DESCRIPTION:
Botulinum toxin type A has been used for hemifacial spasm since 1986. of Botulinum toxin type A can be subcutaneously injected at pretarsal or preseptal portion of orbicularis muscle. Blepharoptosis has been reported less frequently with pretarsal technique, however dry eye was noticed in one patient treated with pretarsal botulinum toxin type A for cosmetic purpose.

ELIGIBILITY:
Inclusion Criteria:

* patient diagnosed with hemifacial spasm

Exclusion Criteria:

* previous history of botulinum toxin treatment for hemifacial spasm
* ocular surface disorders
* tear disorders
* evidence of infection at or around eyelids
* pregnant woman
* other neurologic disease, i.e. OMG
* coagulopathy or treatment with thrombolytic agent
* treatment with aminoglycosides, chloroquine, hydroxychloroquine

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
tear break up time | change from baseline in tear break up time at 12 weeks
  unit of measure; minutes

SECONDARY OUTCOMES:
schirmer's test | change from baseline of schirmer's test at 12 weeks
  units of measurement; millimeters

CONTACTS AND LOCATIONS:
Overall Officials: kitthisak kithaweesin, MD, Principal Investigator — Khon Kaen University
Locations (1):
- Khon Kaen University, Muang, Changwat Khon Kaen, Thailand

REFERENCES:
- [Result] Price J, O'Day J. A comparative study of tear secretion in blepharospasm and hemifacial spasm patients treated with botulinum toxin. J Clin Neuroophthalmol. 1993 Mar;13(1):67-71. PMID 8501266